CLINICAL TRIAL: NCT02768857
Title: A Touch-Observation and Task-based Mirror Therapy Protocol (MTPTOT) to Improve Sensorimotor Control and Functional Capability of Hands for Patients With Peripheral Nerve Injury
Brief Title: Effects of Early Sensory Reeducation Programs Using Mirror Therapy for Patients With Peripheral Nerve Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B-ER-102-389
Record Dates: First submitted 2016-05-05; First posted 2016-05-11 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Sensation Disorders; Motor Deficit; Rehabilitation
MeSH Terms: conditions — Sensation Disorders; Neurologic Manifestations

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Early sensorimotor reeducation intervention (Experimental): The experimental group received 15 minutes of touch-observation and task-based mirror therapy program, followed by 20 minutes of regular hand therapy and 20 minutes of physiotherapy in each treatment session before the returning of the touch of a Semmes-Weinstein monofilament marked 4.31. Once the patients had regained the protective sense (SWM < 4.31), the mirror therapy program was replaced with a discriminative sensory reeducation program. Treatment duration was 12 weeks, at a frequency of three sessions per week.
  Interventions: Behavioral: Sensorimotor reeducation programs
- Traditional sensorimotor reeducation intervention (Active Comparator): The control group received received 15 minutes traditional sensory reeducation program, 20 minutes of regular hand therapy and 20 minutes of physiotherapy in each treatment session before the returning of the touch of a Semmes-Weinstein monofilament marked 4.31. Once the patients had regained the protective sense (SWM < 4.31), the protective sensory reeducation program was replaced with a discriminative sensory reeducation program. Treatment duration was 12 weeks, at a frequency of three sessions per week.
  Interventions: Behavioral: Sensorimotor reeducation programs

INTERVENTIONS:
Behavioral: Sensorimotor reeducation programs

SUMMARY:
This study evaluated the effects of an integrated program of touch-observation and task-based mirror therapy on sensorimotor function in nerve injury patients. Before the return of protective sense (Value of Semmes-Weinstein monofilament test > 4.31), half of the participants received 15 minutes of mirror therapy program, followed by 20 minutes of regular hand therapy and 20 minutes of physiotherapy.While the other half received 15 minutes protective sensory reeducation programs, 20 minutes of regular hand therapy and 20 minutes of physiotherapy in each treatment session. Once the patients had regained the protective sense (Value of Semmes-Weinstein monofilament test < 4.31), the discriminative sensory reeducation program was started for the participants in both groups. The hypothesis was that using the mirror therapy for sensorimotor reeducation in the early phase after nerve repair would yield better results with regard to the returning of sensation, sensorimotor control ability and hand function than using a classical reeducation program alone.

ELIGIBILITY:
Inclusion Criteria:

* median or ulnar nerve injury,
* a combination of nerve and tendon or vascular injury,
* injury sites between the level of mid-palm and elbow, and
* the protective sensation of the hand is lacking or impaired.

Exclusion Criteria:

* patients with deficits in cognition or language comprehension, as well as severe limitations in the range of motion of the upper limbs.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-12; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline result of Semmes-Weinstein monofilament (SWM) test at 12 weeks and 24 weeks | baseline, 12 weeks and 24 weeks
Change from baseline result of Purdue pegboard test at 12 weeks and 24 weeks | baseline, 12 weeks and 24 weeks
Change from baseline result of Minnesota manual dexterity test at 12 weeks and 24 weeks | baseline, 12 weeks and 24 weeks
Change from baseline result of Pinch-holding-up-activity (PHUA) test at 12 weeks and 24 weeks | baseline, 12 weeks and 24 weeks

SECONDARY OUTCOMES:
Change from baseline result of Static two-point discrimination (S2PD) test at 12 weeks and 24 weeks | baseline, 12 weeks and 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng-Kung University Hospital, Tainan, Taiwan, Taiwan